CLINICAL TRIAL: NCT05516394
Title: National Polish Registry of Minimally Invasive Liver Surgery
Acronym: PL-MILS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Jagiellonian University (Other); Ludwik Rydygier Memorial Hospital, Cracow, Poland (Unknown); Regional Oncology Center, Białystok, Poland (Unknown); Medical University of Lublin (Other); Nicolaus Copernicus university Collegium Medicum, Bydgoszcz, Poland (Unknown); Medical University of Łódź (Other)
Responsible Party: Principal Investigator, Wacław Hołówko, Principal Investigator, Medical University of Warsaw
Other Study IDs: AKBE/71/2020
Record Dates: First submitted 2022-08-01; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Liver Tumor
Keywords: laparoscopic liver resection; short-term results; long-term results
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic liver resection — Liver tumors are resected with minimally invasive approach, laparoscopically.

SUMMARY:
After the two consensus meetings on laparoscopic liver resection in Louisville (2008) and in Morioka (2014) minimally invasive approach for liver resection was finally widely established in liver surgery practice. Successively more countries follow laparoscopic liver pioneers and apply laparoscopic liver surgery for everyday practice.

Primary aim of the study is to assess the evolution and diffusion of minimally invasive liver surgery in Poland. Secondly, it will allow to assess the actual short- and long-term results of laparoscopic liver resections and compare it to the international benchmark values.

The National Polish Registry of Minimally Invasive Liver Surgery will include data about all cases of laparoscopic liver resections performed in Poland since the first case in 2010. All surgical departments, where laparoscopic liverresection is regularly performed, will be invited. Data of demography, previous medical history, preoperative assessment, intraoperative and postoperative period, histopathological findings and long-term follow-up will be included in the registry.

This study will be the first national report about diffusion of minimally invasive surgery in Poland.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* underwent laparoscopic liver resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent laparoscopic liver resection in Poland
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 90 days
  Complications in the postoperative period classified by type and their severity according to the Clavien-Dindo grading system

SECONDARY OUTCOMES:
Patient survival | 5 years
Postoperative hospital stay | 1 year
Number of patients scheduled for reoperation after laparoscopic liver resection | 30 days
Number of patients readmitted to hospital after discharge | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Wacław Hołówko, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of General, Transplant and Liver Surgery, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Holowko W, Serednicki W, Bartkowiak M, Wysocki M, Domurat M, Mielko J, Pierscinski S, Hogendorf P, Masior L, Kalinowski P, Wierdak M, Fraczek M, Tarasik A, Wroblewski T, Budzynski A, Pedziwiatr M, Grat M. Early adoption of laparoscopic liver surgery in Poland: a national retrospective cohort study. Int J Surg. 2024 Jan 1;110(1):361-371. doi: 10.1097/JS9.0000000000000840. PMID 37816169